CLINICAL TRIAL: NCT04323722
Title: Impact of Bladder Depletion on Mesorectal Movements During Radiotherapy in Rectal Cancer
Acronym: MESORECT-VV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-2019-15
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer
Keywords: 3D conformal radiotherapy (3DCRT); Intensity-modulated radiotherapy (IMRT); bladder filling; mesorectal movements; filled bladder; empty bladder; cone-beam computerized tomography (CBCT)
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Monocentric, open prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empty bladder (Experimental): Planning CT scan and CBCTs with empty bladder after standard Planning CT scan and CBCTs with filling bladder
  Interventions: Procedure: Empty Bladder planning CT scan and CBCTs

INTERVENTIONS:
Procedure: Empty Bladder planning CT scan and CBCTs — Patient will receive a Planning CT scan, 3 CBCTs on the first week and once a week during radiotherapy treatment with an Empty Bladder

SUMMARY:
This trial is assessing how Bladder filling variations and thus mesorectal movements are less when radiotherapy treatment is received with an empty bladder in rectal cancer

DETAILED DESCRIPTION:
The purpose of this study is to show that the variations of bladder volume and mesorectal movements are less with empty versus filled bladder in rectal cancer.

In this study, patient will be treated with 3D conformal radiotherapy (3D-CRT) radiotherapy with a filled bladder condition, as per standard care, in supine position. A total dose of 45 or 50 Gy in 25 fractions, 5 fractions per week is received.

A Chest, abdomen and pelvis imaging will be performed before treatment start. Patients receive planning CT scan with filled bladder and then with empty bladder on the same day. Only planning CT scan with filled bladder will be used patient treatment.

During radiotherapy treatment, patient will receive CBCTs with filled ans empty bladder on Day 1 ; 2 and 3 on the first week and once a week after.

Multiple parameters will be assessed before treatment (using planning CT scan) and during radiotherapy treatment (CBCTs) in empty ans filled bladder conditions : Bladder volume, mesorectal movements.

A dosimetric study will be performed in Intensity-modulated radiotherapy (IMRT) in empty and filled bladder conditions

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma
* T2 N+ or T3 any N, eligible for radiotherapy or neo-adjuvant radio-chemotherapy treatment in a long course of 25 fractions
* Performance Status less or equal to 2
* Male or female 18 Years and older
* Creatinine clearance greater than or equal to 50ml/min
* Fertile patients must use effective contraception
* Written informed consent
* Patient must be affiliated to a Social Health Insurance

Exclusion Criteria:

* Previous treatment with pelvic radiotherapy
* Chronic inflammatory bowel disease in flare-up.
* Urinary catheterization, urinary diversion or cystectomy
* Hip prosthesis
* History of prostatectomy, or hysterectomy
* Urinary incontinence > 2
* Pregnant or nursing patient
* Persons deprived of their liberty, as well as adults subject to a legal protection measure
* Impossibility to submit to the medical follow-up of this clinical trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Evaluate using imaging techniques and dosimetric analysis the performance of empty versus filled bladder radiotherapy treatment | 3.5 years
  Throughout the radiotherapy treatment, the reproducibility of positioning of the anterior surface of mesorectum will be assessed with empty and filled bladder
Evaluate using imaging techniques and dosimetric analysis the performance of empty versus filled bladder radiotherapy treatment | 3.5 years
  Throughout the radiotherapy treatment, the reliability of positioning of the anterior surface of mesorectum will be assessed with empty and filled bladder

SECONDARY OUTCOMES:
Evaluate mesorectal movements during radiotherapy in empty versus filled bladder | 3.5 years
  Compare mesorectal movements during radiotherapy treatment compared to the planning CT scan in the case of a filled versus an empty bladder
Evaluate changes in bladder volume during radiotherapy in empty versus filled bladder | 3.5 years
  Compare changes in bladder volume during treatment versus planning CT scan for filled bladder versus empty bladder
IMRT (Intensity-Modulated Radiotherapy) dosimetric study in patients with filled or empty bladder | 3.5 years
  Compare and validate (in silico on planning CT scan) the compliance with dose constraints to organs-at-risk in patients with filled or empty bladder in IMRT

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut de Cacerologie de l'ouest - site Paul Papin, Angers
  - ICO René Gauducheau, Saint-Herblain